CLINICAL TRIAL: NCT04748432
Title: Lipid Kinetics of Patients With Nonfermenting Gram-Negative Bacterial Ventilator-Associated Pneumonia
Brief Title: Lipid Kinetics of Patients With Pneumonia
Status: Completed | Type: Observational
Sponsor: Konya Numune Hospital (Other Government)
Responsible Party: Principal Investigator, Omur ILBAN, Principal investigator, Konya Numune Hospital
Other Study IDs: omurilban
Record Dates: First submitted 2021-02-03; First posted 2021-02-10 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Gram-negative Bacteria; Lipid Metabolism; Nosocomial Infections
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Multi-drug resistant group (MDR): Patients with resistant NFGNB isolate as MDR group
- Non-Multi-drug resistant group (Non-MDR): Patients with sensitive NFGNB isolate as Non-MDR group
- Control group (Control): Patients without suspicion of VAP and other signs of nosocomial infection as the control group

SUMMARY:
Nonfermenting Gram-Negative Bacilli (NFGNB) are aerobic, non-motile, non-lactose fermenting, oxidase-negative, catalase-positive coccobacilli that pose a serious threat to critically ill patients. Primarily Pseudomonas aeruginosa (PA) and Acinetobacter baumannii (AB), are NFGNB which are potential multi-drug resistant (MDR) pathogens that are related to ventilator-associated pneumonia (VAP). In Nonfermenting Gram-Negative Bacilli (NFGNB) infections, which are potential multi-drug resistant (MDR) pathogens, pathogenesis is determined not only by bacterial virulence factors but more importantly by the interaction between bacteria and the host immune system. Thanks to their direct immunomodulatory properties, lipoproteins and lipids bind and neutralise toxic bacterial substances. During the acute phase response and inflammation, HDL presents significant structural and functional changes. This study was planned to evaluate the relationship between the changes of the serum lipid metabolism and other inflammation markers with the antimicrobial resistance status and the results in NFGNB VAP patients. Also, we aimed to investigate whether there is a difference in the clinical characteristics of the patients depending on the resistance profile of NFGNB.

DETAILED DESCRIPTION:
This prospective study was performed in adult intensive care unit (ICU) patients. They were intubated endotracheally and received mechanical ventilation (MV) treatment for at least 48 hours in Konya Numune Hospital ICU, which has 42 surgery and medicine beds. The study was conducted between May 2019 and December 2020 and approved by the Ethics Committee of Necmettin Erbakan University Medical School. Informed consents were obtained from the patients who participated in the study or from their relatives. The characteristics of the patients and the sequential changes of the inflammatory response including the lipid profile were recorded.

ELIGIBILITY:
Inclusion Criteria:

* ICU Patients of 18 years of age and above, with clinical suspicion of VAP as defined in the American Thoracic Society (ATS) guidelines and a simplified version of Clinical Pulmonary Infection Score (CPIS)> 6, with significant NFGNB growth in respiratory cultures and with no signs and symptoms of infection at the time of admission, were included in the study.

Exclusion Criteria:

* Patients with chronic inflammatory disease, hepatic dysfunction, active tuberculosis, malignancy, malnutrition, severe immunosuppression (i.e., neutropenia, HIV positive, organ transplant, having received immunosuppressants or used ≥ 20 mg/day prednisone for two or more weeks in the preceding three months), those that within 72 hours since being included in the study had any extrapulmonary infection other than VAP, as well as those whose respiratory cultures presented bacterial agents other than NFGNB and fungal agents were not included in the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients who were intubated endotracheally and received mechanical ventilation treatment for at least 48 hours in ICU.
Sampling Method: Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2019-05-25 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Serum lipid metabolism | 18 months
  The relationship between the changes of the serum lipid metabolism including total cholesterol, high-density lipoprotein cholesterol, low-density lipoprotein cholesterol and triglycerides with the antimicrobial resistance status and the results in NFGNB VAP patients

SECONDARY OUTCOMES:
Clinical outcome | 18 months
  The secondary outcome were the 30-day mortality rate of the patients depending on the resistance profile of NFGNB

CONTACTS AND LOCATIONS:
Overall Officials: Omur ILBAN, MD, Principal Investigator — Konya Numune Hospital, Department of Intensive Care
Locations (1):
- Konya Numune Hospital, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided